CLINICAL TRIAL: NCT01645280
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Study Evaluating the Efficacy and Safety of Ustekinumab (STELARA®) and CNTO 1959 Administered Subcutaneously in Subjects With Active Rheumatoid Arthritis Despite Concomitant Methotrexate Therapy
Brief Title: A Study of the Effectiveness and Safety of Ustekinumab (STELARA) and CNTO 1959 Administered Under the Skin of Patients With Active Rheumatoid Arthritis, Despite Existing Methotrexate Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100736; CNTO1275ARA2001 (Other: Janssen Research & Development, LLC); 2011-001122-18 (EudraCT Number)
Record Dates: First submitted 2012-06-06; First posted 2012-07-20 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: Active rheumatoid arthritis; Ustekinumab; STELARA; CNTO 1959
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Ustekinumab; guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Placebo Comparator)
  Interventions: Drug: Placebo + methotrexate (MTX) (Group 1)
- Group 2 (Experimental)
  Interventions: Drug: Ustekinumab + MTX (Group 2)
- Group 3 (Experimental)
  Interventions: Drug: Ustekinumab + MTX (Group 3)
- Group 4 (Experimental)
  Interventions: Drug: CNTO 1959 + MTX (Group 4)
- Group 5 (Experimental)
  Interventions: Drug: CNTO 1959 + MTX (Group 5)

INTERVENTIONS:
Drug: Placebo + methotrexate (MTX) (Group 1) — Placebo: form = solution for injection, route = subcutaneous use, at Weeks 0, 4, then every 8 weeks (Weeks 12, 20, and 28) + MTX (pre-study dose)
  Arms: Group 1
Drug: Ustekinumab + MTX (Group 2) — Ustekinumab: type = exact number, unit = mg, number = 90, form = solution for injection, route = subcutaneous use, at Weeks 0, 4, then every 8 weeks (Weeks 12, 20, and 28) + MTX (pre-study dose)
  Arms: Group 2
Drug: Ustekinumab + MTX (Group 3) — Ustekinumab: type = exact number, unit = mg, number = 90, form = solution for injection, route = subcutaneous use, at Weeks 0, 4, then every 12 weeks (Weeks 16 and 28) + MTX (pre-study dose)
  Arms: Group 3
Drug: CNTO 1959 + MTX (Group 4) — CNTO 1959: type = exact number, unit = mg, number = 200, form = powder for solution for injection, route = subcutaneous use, at Weeks 0, 4, then every 8 weeks (Weeks 12, 20, and 28) + MTX (pre-study dose)
  Arms: Group 4
Drug: CNTO 1959 + MTX (Group 5) — CNTO 1959: type = exact number, unit = mg, number = 50, form = powder for solution for injection, route = subcutaneous use, at Weeks 0, 4, then every 8 weeks (Weeks 12, 20, and 28)+ MTX (pre-study dose)
  Arms: Group 5

SUMMARY:
The purpose of this study is to evaluate the efficacy of ustekinumab and CNTO 1959 in reducing the signs and symptoms of disease in patients with active rheumatoid arthritis (RA) despite concomitant methotrexate (MTX) therapy and to evaluate the safety of ustekinumab and CNTO 1959 in this population.

DETAILED DESCRIPTION:
This is a randomized (patients assigned to treatment by chance), double-blind (study personnel and patients will not know what treatment is being assigned to patients), multicenter, placebo-controlled (a placebo is a treatment identical in appearance to the study agent, but containing no active ingredient), dose-ranging study. Approximately 250 patients will be randomly assigned to 1 of 5 treatment groups. The maximum length of study participation is 54 weeks, including a 6-week screening period. The end of the study will be the last follow-up visit of the last patient. Study visits and evaluations will occur, and patient safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have had RA for at least 6 months prior to screening
* Have a diagnosis of RA according to the revised 1987 criteria of the American Rheumatism Association - Be positive for either anti-cyclic citrullinated peptide antibody or rheumatoid factor in serum at screening
* Have been treated with and tolerated MTX for at least 6 months prior to screening, and have a MTX dose of >= 10 mg and <= 25 mg per week and stable for at least 12 weeks prior to first administration of study agent
* Have active RA, defined as persistent disease activity with both of the following criteria: at least 6 swollen and 6 tender joints at the time of screening and baseline; serum C-reactive protein (CRP) >= 0.80 mg/dL at screening. The investigator may consider the patient eligible if the CRP value is at least 0.80 mg/dL in a single repeat testing during the screening period
* If using oral corticosteroids, must be on a stable dose of <= 10 mg/day of prednisone or an equipotent dose of another oral corticosteroid for at least 2 weeks prior to the first administration of study agent. If not using corticosteroids at Week 0, the patient must not have received oral corticosteroids for at least 2 weeks prior to the first administration of study agent
* If using nonsteroidal anti-inflammatory drugs (NSAIDs) or other analgesics regularly for RA, the patient must have been on a stable dose for at least 2 weeks prior to the first administration of study agent. If not using NSAIDs or other analgesics for RA at Week 0, the patient must have not received NSAIDs or other analgesics for RA for at least 2 weeks prior to the first administration of study agent

Exclusion Criteria:

* Has other inflammatory diseases, including but not limited to psoriatic arthritis, ankylosing spondylitis (AS), systemic lupus erythematosus, or Lyme disease, that might confound the evaluation of the benefit of study agent therapy
* Has current signs or symptoms of liver insufficiency or cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, psychiatric, or metabolic disturbances that are severe, progressive, or uncontrolled
* Has any known malignancy or history of malignancy (with the exception of basal cell carcinoma, squamous cell carcinoma in situ of the skin, or cervical carcinoma in situ that has been treated with no evidence of recurrence, or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years prior to the first administration of study agent)
* Has a history of lymphoproliferative disease, including lymphoma, or signs suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location, or clinically significant splenomegaly
* Has known allergies, hypersensitivity, or intolerance to ustekinumab or CNTO 1959 or its inactive ingredients
* Has ever received any approved or investigational biologic agent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (47):
- United States (3):
  - Palm Harbor, Florida
  - Rock Island, Illinois
  - St Louis, Missouri
- Argentina (3):
  - Buenos Aires
  - San Juan
  - San Miguel de Tucumán
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Osorno, Chile
- Colombia (5):
  - Bogotá
  - Bucaramanga
  - Cali
  - Chía
  - Medellín
- Czechia (3):
  - Hlučín
  - Kladno
  - Uherské Hradiště
- Hungary (5):
  - Budapest
  - Gödöllő
  - Székesfehérvár
  - Szombathely
  - Veszprém
- Poland (7):
  - Bialystok
  - Elblag
  - Krakow
  - Poznan
  - Sopot
  - Sosnowiec
  - Warsaw
- Russia (9):
  - Kazan'
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Saint Petersburg
  - Saratov
  - Ufa
  - Ulyanovsk
  - Yaroslavl
- Singapore, Singapore
- Ukraine (8):
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Simferopol
  - Ternopil
  - Uzhhorod
  - Vinnitsa

REFERENCES:
- [Derived] Smolen JS, Agarwal SK, Ilivanova E, Xu XL, Miao Y, Zhuang Y, Nnane I, Radziszewski W, Greenspan A, Beutler A, Baker D. A randomised phase II study evaluating the efficacy and safety of subcutaneously administered ustekinumab and guselkumab in patients with active rheumatoid arthritis despite treatment with methotrexate. Ann Rheum Dis. 2017 May;76(5):831-839. doi: 10.1136/annrheumdis-2016-209831. Epub 2017 Jan 13. PMID 28087506

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 274 subjects were enrolled into the study and 273 were treated. One participant in the Ustekinumab 90 milligram (mg) every 8 weeks group did not receive the treatment due to an adverse event before dosing.
Groups:
- Placebo: Participants randomized to receive matching placebo subcutaneously at Week 0, 4 and then every 8 weeks (Week 12, 20 and 28) along with methotrexate. 16 participants in placebo group early escaped to receive the study drug Ustekinmab.
- Ustekinumab 90 mg Every 8 Weeks: Participants randomized to receive ustekinumab 90 milligram (mg) subcutaneously at Week 0, 4 and then every 8 weeks (Week 12, 20 and 28) along with methotrexate.
- Ustekinumab 90 mg Every 12 Weeks: Participants randomized to receive ustekinumab 90 milligram (mg) subcutaneously at Week 0, 4 and then every 12 weeks (Week 16 and 28) along with methotrexate.
- CNTO1959 200 mg Every 8 Weeks: Participants randomized to receive CNTO1959 200 mg subcutaneously at Week 0, 4 and then every 8 weeks (Week 12, 20 and 28) along with methotrexate.
- CNTO1959 50 mg Every 8 Weeks: Participants randomized to receive CNTO1959 50 mg subcutaneously at Week 0, 4 and then every 8 weeks (Week 12, 20 and 28) along with methotrexate.
Period: Overall Study
Arm/Group | Placebo | Ustekinumab 90 mg Every 8 Weeks | Ustekinumab 90 mg Every 12 Weeks | CNTO1959 200 mg Every 8 Weeks | CNTO1959 50 mg Every 8 Weeks
Started | 55 (16 participants in placebo group early escaped to receive Ustekinmab; included in safety population.) | 54 | 55 | 54 | 55
Completed | 49 | 51 | 49 | 48 | 47
Not Completed | 6 | 3 | 6 | 6 | 8
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 2 | 4 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1
Not completed — Other | 1 | 1 | 2 | 0 | 0
Not completed — Treatment not completed/Completed f/u | 1 | 1 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ustekinumab 90 mg Every 8 Weeks | Ustekinumab 90 mg Every 12 Weeks | CNTO1959 200 mg Every 8 Weeks | CNTO1959 50 mg Every 8 Weeks | Total
Number analyzed (Participants) | 55 | 55 | 55 | 54 | 55 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (10.57) | 50.8 (13.01) | 51.4 (13.59) | 54.6 (11.34) | 49.9 (12.85) | 51.5 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 47 | 42 | 45 | 228
  Male | 7 | 9 | 8 | 12 | 10 | 46
Region of Enrollment [Number; unit: participants]
  Argentina | 1 | 5 | 6 | 5 | 6 | 23
  Bulgaria | 2 | 2 | 2 | 2 | 1 | 9
  CZ Rep | 0 | 0 | 1 | 0 | 0 | 1
  Chile | 1 | 1 | 1 | 1 | 2 | 6
  Colombia | 10 | 9 | 8 | 6 | 10 | 43
  Hungary | 6 | 5 | 2 | 4 | 3 | 20
  Poland | 5 | 8 | 6 | 7 | 9 | 35
  Russia | 20 | 15 | 18 | 19 | 14 | 86
  Singapore | 1 | 1 | 0 | 2 | 0 | 4
  USA | 0 | 0 | 1 | 0 | 0 | 1
  Ukraine | 9 | 9 | 10 | 8 | 10 | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology 20 (ACR 20) Response at Week 28
Description: The ACR 20 responders are participants with at least 20 percent (%) improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) patient's assessment of arthritis pain-visual analog scale, 2) patient's global assessment of disease activity-visual analog scale, 3) physician's global assessment of disease activity-visual analog scale, 4) patient's assessment of physical function as measured by health assessment questionnaire-disability index (HAQ-Di), 5) C-reactive protein (CRP).
Time Frame: Week 28
Population: The intent-to-treat (ITT) population included all randomized participants. For early escape, data at or prior to Week 16 were carried forward through Week 28.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ustekinumab 90 mg Every 8 Weeks | Ustekinumab 90 mg Every 12 Weeks | CNTO1959 200 mg Every 8 Weeks | CNTO1959 50 mg Every 8 Weeks
Number analyzed (Participants) | 55 | 55 | 55 | 54 | 55
percentage of participants | 40.0 | 52.7 | 54.5 | 44.4 | 38.2
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 90 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.184, Cochran-Mantel-Haenszel; Screening CRP level (>= 1.50 mg/dL; < 1.50 mg/dL) was used as stratification factors
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg Every 12 Weeks; Test type: Superiority or Other; p = 0.130, Cochran-Mantel-Haenszel; Screening CRP level (>= 1.50 mg/dL; < 1.50 mg/dL) was used as stratification factors
Statistical Analysis 3: Comparison: Placebo vs CNTO1959 200 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.642, Cochran-Mantel-Haenszel; Screening CRP level (>= 1.50 mg/dL; < 1.50 mg/dL) was used as stratification factors
Statistical Analysis 4: Comparison: Placebo vs CNTO1959 50 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.832, Cochran-Mantel-Haenszel; Screening CRP level (>= 1.50 mg/dL; < 1.50 mg/dL) was used as stratification factors

2. Secondary Outcome: Change From Baseline in Disease Activity Index Score 28 (DAS28; Using C-reactive Protein [CRP]) Score at Week 28
Description: The DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, CRP (mG/L) and patient's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: From Baseline to Week 28
Population: The modified-ITT population included participants who received at least 1 (partial or complete) dose of study agent. For early escape, data at or prior to Week 16 were carried forward through Week 28.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Ustekinumab 90 mg Every 8 Weeks | Ustekinumab 90 mg Every 12 Weeks | CNTO1959 200 mg Every 8 Weeks | CNTO1959 50 mg Every 8 Weeks
Number analyzed (Participants) | 55 | 54 | 55 | 54 | 55
units on scale | -0.94 (0.174) | -1.52 (0.185) | -1.49 (0.183) | -1.21 (0.170) | 6.07 (0.821)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 90 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.019, ANCOVA; Treatment, screening CRP level (>=1.50 mg/dL, <1.50mg/dL) and baseline score as covariates
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg Every 12 Weeks; Test type: Superiority or Other; p = 0.025, ANCOVA; Treatment, screening CRP level (>=1.50 mg/dL, <1.50mg/dL) and baseline score as covariates
Statistical Analysis 3: Comparison: Placebo vs CNTO1959 200 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.248, ANCOVA; Treatment, screening CRP level (>=1.50 mg/dL, <1.50mg/dL) and baseline score as covariates
Statistical Analysis 4: Comparison: Placebo vs CNTO1959 50 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.045, ANCOVA; Treatment, screening CRP level (>=1.50 mg/dL, <1.50mg/dL) and baseline score as covariates

3. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20 (ACR 20) Response at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: The m-ITT population included participants who received at least 1 (partial or complete) dose of study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ustekinumab 90 mg Every 8 Weeks | Ustekinumab 90 mg Every 12 Weeks | CNTO1959 200 mg Every 8 Weeks | CNTO1959 50 mg Every 8 Weeks
Number analyzed (Participants) | 55 | 54 | 55 | 54 | 55
percentage of participants | 29.1 | 37.0 | 34.5 | 33.3 | 20.0
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 90 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.381, Cochran-Mantel-Haenszel; Screening CRP level (>= 1.50 mg/dL; < 1.50 mg/dL) was used as stratification factors
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg Every 12 Weeks; Test type: Superiority or Other; p = 0.543, Cochran-Mantel-Haenszel; Screening CRP level (>= 1.50 mg/dL; < 1.50 mg/dL) was used as stratification factors
Statistical Analysis 3: Comparison: Placebo vs CNTO1959 200 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.629, Cochran-Mantel-Haenszel; Screening CRP level (>= 1.50 mg/dL; < 1.50 mg/dL) was used as stratification factors
Statistical Analysis 4: Comparison: Placebo vs CNTO1959 50 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.273, Cochran-Mantel-Haenszel; Screening CRP level (>= 1.50 mg/dL; < 1.50 mg/dL) was used as stratification factors

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Week 28
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI): participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline and Week 28
Population: The m-ITT included participants who received at least 1 (partial or complete) dose of study agent. For early escape, data at or prior to Week 16 were carried forward through Week 28.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | Ustekinumab 90 mg Every 8 Weeks | Ustekinumab 90 mg Every 12 Weeks | CNTO1959 200 mg Every 8 Weeks | CNTO1959 50 mg Every 8 Weeks
Number analyzed (Participants) | 55 | 54 | 55 | 54 | 55
units on scale | -0.30 (0.074) | -0.48 (0.072) | -0.44 (0.071) | -0.41 (0.075) | -0.39 (0.076)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 90 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.060, ANCOVA; Treatment, screening CRP level (>=1.50 mg/dL, <1.50mg/dL) and baseline score as covariates
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg Every 12 Weeks; Test type: Superiority or Other; p = 0.134, ANCOVA; Treatment, screening CRP level (>=1.50 mg/dL, <1.50mg/dL) and baseline score as covariates
Statistical Analysis 3: Comparison: Placebo vs CNTO1959 200 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.280, ANCOVA; Treatment, screening CRP level (>=1.50 mg/dL, <1.50mg/dL) and baseline score as covariates
Statistical Analysis 4: Comparison: Placebo vs CNTO1959 50 mg Every 8 Weeks; Test type: Superiority or Other; p = 0.345, ANCOVA; Treatment, screening CRP level (>=1.50 mg/dL, <1.50mg/dL) and baseline score as covariates

ADVERSE EVENTS:
Time Frame: Week 0 to 48
Description: Safety population included all participants who received at least 1 dose of study drug.
Groups:
- Placebo (Early Escape): Participants who early escaped at Week 16 and received ustekinumab 90 milligram (mg) subcutaneously at Week 16, 20 and 28 along with methotrexate.
Arm/Group | Placebo | Placebo (Early Escape) | Ustekinumab 90 mg Every 8 Weeks | Ustekinumab 90 mg Every 12 Weeks | CNTO1959 200 mg Every 8 Weeks | CNTO1959 50 mg Every 8 Weeks
Serious Adverse Events (participants affected / at risk) | 3/55 | 1/16 | 4/54 | 3/55 | 3/54 | 0/55
Other Adverse Events (participants affected / at risk) | 13/55 | 6/16 | 15/54 | 15/55 | 18/54 | 14/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Placebo (Early Escape) (N=16) | Ustekinumab 90 mg Every 8 Weeks (N=54) | Ustekinumab 90 mg Every 12 Weeks (N=55) | CNTO1959 200 mg Every 8 Weeks (N=54) | CNTO1959 50 mg Every 8 Weeks (N=55)
Angina Unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Breast Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Placebo (Early Escape) (N=16) | Ustekinumab 90 mg Every 8 Weeks (N=54) | Ustekinumab 90 mg Every 12 Weeks (N=55) | CNTO1959 200 mg Every 8 Weeks (N=54) | CNTO1959 50 mg Every 8 Weeks (N=55)
Influenza (Infections and infestations) | 3 | 0 | 1 | 3 | 3 | 3
Nasopharyngitis (Infections and infestations) | 3 | 1 | 5 | 4 | 4 | 3
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 5 | 4 | 2
Headache (Nervous system disorders) | 3 | 1 | 2 | 5 | 3 | 2
Hypertension (Vascular disorders) | 3 | 1 | 4 | 2 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 3 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 2 | 4 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 2 | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.